CLINICAL TRIAL: NCT03828084
Title: An Open-Label, Randomized, Single-Dose, Four-Way Crossover, Bioavailability Study of Three Formulations of Decitabine/Tetrahydrouridine (THU) Combination Modified Release Capsules (5 mg/250 mg) in Healthy and Fasting Adults
Brief Title: Randomized, Single-dose, Crossover Study of 4 Decitabine and Tetrahydrouridine (EPI01) Formulations in Healthy Subjects
Acronym: EPI01
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EpiDestiny, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: EPI-01-CP.001
Record Dates: First submitted 2019-01-31; First posted 2019-02-04 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Healthy
MeSH Terms: interventions — Decitabine; Tetrahydrouridine

STUDY DESIGN:
Intervention Model Description: Four-way crossover, single dose with a 7 days washout period in between periods
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Formulation A (Experimental): 3 test capsules of combination decitabine/THU (5 mg/250 mg per capsule; Formulation A) given as a single oral dose with approximately 240 mL (8 fluid ounces) of ambient temperature water.
  Interventions: Drug: Decitabine
- Formulation B (Experimental): 3 test capsules of combination decitabine/THU (5 mg/250 mg per capsule; Formulation B) given as a single oral dose with approximately 240 mL (8 fluid ounces) of ambient temperature water.
  Interventions: Drug: Decitabine
- Formulation C (Experimental): 3 test capsules of combination decitabine/THU (5 mg/250 mg per capsule; Formulation C) given as a single oral dose with approximately 240 mL (8 fluid ounces) of ambient temperature water.
  Interventions: Drug: Decitabine
- Reference Formulation (Active Comparator): 3 capsules of THU (250 mg per capsule) given as a single oral dose with approximately 240 mL of ambient temperature water, followed by a single oral dose of 3 capsules of decitabine (5 mg per capsule) given 1 hour later with approximately 240 mL of ambient temperature water.
  Interventions: Drug: Decitabine

INTERVENTIONS:
Drug: Decitabine — Combination drugs containing decitabine and tetrahydrouridine
  Other Names: Tetrahydrouridine

SUMMARY:
To study the pharmacokinetic profiles of decitabine and tetrahydrouridine (THU) from 3 modified release formulations in healthy subjects.

DETAILED DESCRIPTION:
This is an open-label, randomized, single-dose per period, four-period, crossover study to evaluate relative bioavailability of decitabine in three newly formulated THU and decitabine combination capsules in comparison to 3 capsules of THU followed 1 hour later by 3 capsules of decitabine.

ELIGIBILITY:
Inclusion Criteria:

* Must understand and voluntarily sign a written ICF prior to any study related procedures being performed and be able to adhere to restrictions and examination schedules.
* Must be able to communicate with the investigator, and to understand and comply with the requirements of the study.
* Healthy male volunteers from any race between 18 to 50 years of age (inclusive), and in good health as determined by past medical history, physical examination, vital signs, ECG, and laboratory tests at screening.
* Must have a body mass index (BMI) between 18 and 30 kg/m2 (inclusive) and a weight between 60 and 100 kg (132 to 220 lb), inclusive, at screening.
* Subject's clinical laboratory test results have no clinically significant findings, in the opinion of the Investigator.
* Vital signs (systolic and diastolic blood pressure and pulse rate) will be assessed in the supine position after the subject has rested for at least 5 minutes. At screening, the potential subject must be afebrile, with a systolic blood pressure between 90 and 140 mmHg (inclusive), diastolic blood pressure between 60 and 90 mmHg (inclusive), and pulse rate between 50 and 100 bpm (inclusive). Vital signs criteria at each check-in and the pre-dose measurements will be at the Investigator's discretion.
* Subjects must be free of any clinically significant disease that would interfere with the study evaluations.
* Subjects (including those who have had a documented vasectomy) must be using a double-barrier local contraception (i.e., spermicidal gel plus condom) when engaging in sexual activity with women of childbearing potential while on study medication and for 28 days after the last dose of study medication.
* Subjects must refrain from sperm donations while on study drug, for the entire duration of the study, and for 28 days after the last dose of study drug.

Exclusion Criteria:

* History or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, oncologic, or psychiatric disease or any other condition, including the presence of laboratory abnormalities, that, in the opinion of the Investigator, would jeopardize the safety of the subject or the validity of the study results.
* Any serious medical condition, clinically significant laboratory abnormality, or psychiatric illness that would prevent the subject from signing the ICF.
* Recent history within 3 years of any clinically significant neurological, gastrointestinal, renal, hepatic, cardiovascular, psychological, pulmonary, metabolic, endocrine, hematological or other major disorders.
* Used any prescribed systemic or topical medication within 30 days of the first dose administration.
* Used any non-prescribed systemic (including herbal medicines, e.g. St. John's Wort) or topical medication within 7 days of the first dose administration (with the exception of vitamin/mineral supplements)
* Subjects who have any surgical or medical conditions possibly affecting drug absorption, distribution, metabolism and excretion (ADME).
* Exposed to an investigational drug (new chemical entity) within 90 days preceding the first dose administration or currently enrolled in any investigational trials.
* Donated blood or plasma within 8 weeks preceding the first dose administration.
* History of multiple drug allergies.
* Any clinically significant allergic disease (excluding nonactive hay fever).
* History of drug abuse of at least 2 years prior to dosing, or positive drug screening test due to illicit drugs.
* History of alcohol abuse of at least 2 years prior to dosing, or positive alcohol screen.
* Smokers or users of other tobacco products (e.g., chewing tobacco, or those using nicotine-containing products (i.e., patches, gum) in the 3 months prior to screening, or positive urine cotinine test.
* Known to have serum hepatitis or known to be a carrier of the hepatitis B surface antigen (HBsAg) or hepatitis C antibody, or tests positive for HIV (human immunodeficiency virus) antibodies at screening.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-04-03 (Actual); Primary Completion 2019-05-02 (Actual); Study Completion 2019-05-03 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of Decitabine | 24 hours
  Area under the concentration-time curve (AUC) from time of dosing to the last quantifiable concentration of Decitabine
Decitabine plasma concentration | 24 hours
  Maximum concentration (Cmax) of Decitabine in plasma
Pharmacokinetics of Tetrahydrouridine | 24 hours
  Area under the concentration-time curve (AUC) from time of dosing to the last quantifiable concentration of THU

SECONDARY OUTCOMES:
Safety of Decitabine and Tetrahydrouridine | 24 hours
  Safety of single dose as measured by adverse event reporting

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia A Zamora, MD, Principal Investigator — Worldwide Clinical Trials Early Phase Services, LLC
Locations (1):
- Worldwide Clinical Trial, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

REFERENCES:
- See also: To participate in a Worldwide clinical trial — https://www.worldwide.com/participate-in-a-study/